CLINICAL TRIAL: NCT00884130
Title: Cost Effectiveness of Laparoscopic Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Collaborators: Minimal Access Therapy Training Unit (Other); Ethicon Endo-Surgery (Europe) GmbH (Industry)
Responsible Party: Alison Sawyer, Postgraduate Medical School, University of Surrey
Other Study IDs: 05/Q1909/74
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Colorectal Surgery
Keywords: Laparoscopy; Colorectal surgery; Quality of life; economic analysis; Patients undergoing laparoscopic colorectal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laparoscopic: Patients having a laparoscopic colorectal resection
  Interventions: Procedure: laparoscopic colorectal resection
- Open: Patients having an open colorectal resection
  Interventions: Procedure: open colorectal resection

INTERVENTIONS:
Procedure: laparoscopic colorectal resection
  Groups: Laparoscopic
Procedure: open colorectal resection
  Groups: Open

SUMMARY:
Hypothesis: The total costs of laparoscopic colorectal surgery are less than those of open surgery.

Secondary hypothesis: Patients quality of life is higher following laparoscopic surgery, as compared to open colorectal surgery.

Research objectives:

1. To estimate the cost implications and clinical benefits of incorporating laparoscopic colorectal surgery into routine clinical practice.
2. To examine whether the increased operative costs of laparoscopic surgery are compensated for by a faster recovery, shorter duration of hospital stay, and a reduction in late complications, as compared to open surgery.
3. To investigate whether there are differences in quality of life following laparoscopic colorectal surgery as compared to open surgery.

Lay summary:

Patients needing an operation for a bowel problem have traditionally had an open operation with an incision on the abdomen, and this is the type of operation that is currently performed in the majority of cases in the United Kingdom today (over 90%). Laparoscopic (or keyhole) surgery has been introduced into bowel surgery, but is currently not widely performed. This is because thus far there have been no clear-cut benefits demonstrated with this technique and the perceived costs are higher than an open operation. The investigators aim to evaluate both of these issues.

ELIGIBILITY:
Inclusion Criteria:

* All patients having a colorectal resection, including benign and malignant tumours, inflammatory bowel disease, diverticular disease, and endometriosis

Exclusion Criteria:

* Children
* Emergency procedures
* Patients unable to consent, unable to complete a quality of life diary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients requiring a colorectal resection between January 2006 and August 2007 at The Royal Surrey County Hospital, UK.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The cost effectiveness of laparoscopic colorectal surgery | 6 weeks

SECONDARY OUTCOMES:
Costs of laparoscopic and open colorectal surgery | 6 weeks
Quality of life of patients having laparoscopic and open colorectal surgery | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henry m Dowson, MBBS FRCS, Principal Investigator — Minimal Access Therapy Training Unit; Timothy Rockall, MBBS FRCS, Study Chair — Minimal Access Therapy Training Unit
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom